CLINICAL TRIAL: NCT00746616
Title: Durom(R) Hip Resurfacing System Multicenter Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-100; G060120/S6
Record Dates: First submitted 2008-09-02; First posted 2008-09-04 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: Advanced Hip Disease
Keywords: Total Hip Arthroplasty,; Acetabular Cup,; Hip Resurfacing; Young,; active; patients
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Hip resurfacing devices in the young, active patient with advanced hip disease instead of traditional total hip arthroplasty.
  Interventions: Device: Durom Hip Resurfacing System

INTERVENTIONS:
Device: Durom Hip Resurfacing System — Hip resurfacing devices in the young, active patient with advanced hip disease instead of traditional total hip arthroplasty.
  Other Names: Hip Reserfacing

SUMMARY:
The purpose of the study is to gather clinical information on the safety and efficacy of the resurfacing devices in the young, active patient with advanced hip disease. Study enrollment has been temporarily suspended due to a change in the surgical technique.

DETAILED DESCRIPTION:
Safety will be evaluated based on the frequency and incidence of any device related adverse events or unanticipated adverse device events. The efficacy will be measured by comparing the overall functional performance based on the Harris Hip Score, implant survivorship, and radiographic parameters, including radiolucencies, osteolysis, stem subsidence, cup migration, and change in cup angle and a change in the femoral shaft angle.

ELIGIBILITY:
Inclusion Criteria:

* Patient selection without bias to race or gender
* Patient is greater than or equal to 18 and less than or equal to 65 years of age.
* Female patients only:

  * actively practicing a contraceptive method, or
  * surgically sterilized, or
  * post-menopausal
* Pre-operative Harris Hip Score less than or equal to 70.
* Primary surgical hip candidate, suffering from hip pain and/or disability due to degenerative joint disease (inflammatory or non-inflammatory), based on physical examination and history, including the following diagnosis:

  * non-inflammatory degenerative joint disease (NIDJD), e.g. avascular necrosis or osteoarthritis
  * inflammatory joint disease (IJD), e.g. rheumatoid arthritis
* Patient is willing and able to cooperate in prescribed post-operative therapy.
* Patient is willing and able to complete scheduled follow-up evaluations as described in the Informed Consent.
* Patient has participated in the Informed Consent process and has signed and IRB approved Informed Consent.

Exclusion Criteria:

* Patient with an acute, chronic, local or systemic infection.
* Patient who is skeletally immature.
* Patient with a severe muscular, neural or vascular disease that endangers the involved extremity.
* Patient with an insufficient acetabular or femoral bone stock in which good anchorage of the implants are unlikely or impossible, including but not limited to:

  * patient with severe osteopenia
  * patients with a family history of severe osteoporosis or osteopenia
  * patients with osteonecrosis or avascular necrosis (AVN) with > 50% involvement of the femoral head (regardless of FICAT grade)
  * patients with multiple cysts of the femoral head > 1cm
* Patient with total or partial absence of the muscular of ligamentous apparatus.
* Patient has known moderate to severe renal insufficiency.
* Patient with a known clinical condition which may interfere with patient outcome, including but not limited to:

  * immuno-compromised conditions (AIDS),
  * organ transplant recipient,
  * high doses of corticosteroids etc
* Patient who is severely overweight (BMI >40)
* Operative (ipsilateral) Hip: Patient has a total prosthetic hip replacement device, surface arthroplasty or endoprosthesis.
* Contralateral Hip: Patient has had hip replacement, surface arthroplasty or endoprosthesis, within the past 12 months, unless already enrolled in this investigational study.
* Patient who is:

  * a prisoner
  * mentally incompetent
  * a known alcohol or drug abuser
  * anticipated to be non-compliant
* Patient who has participated in a study of any other investigational device (drug, device or biologic) within the past 12 months. Exception: previous enrollment in the Durom Hip Resurfacing System clinical study.
* Patient has a known allergy to one of the constituents of the implant, e.g. cobalt, chromium, nickel, etc.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-06; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Device Survival | All post-op visits until last patient enrolled reaches 2 year follow-up

SECONDARY OUTCOMES:
Efficacy | 6 month post-op and annually until last patient reaches 2 year follow-up

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Colorado Joint Replacement, Denver, Colorado
  - Syracuse Orthopedic Specialists, De Witt, New York
  - Eastern Oklahoma Orthopedic Center, Tulsa, Oklahoma
  - PENN Orthopedics, Philadelphia, Pennsylvania
  - Texas Hip and Knee, Fort Worth, Texas